CLINICAL TRIAL: NCT05311436
Title: Nutri-CAP: Nutrition for Children, Adolescent Girls, and Pregnant Women in Slums of Dhaka City
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Global Affairs Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-21082
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Gestational Weight Gain; Diet, Food, and Nutrition; Undernutrition; Health Behavior
MeSH Terms: conditions — Gestational Weight Gain; Malnutrition; Health Behavior | interventions — Gravidity; Iron; Folic Acid; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): 1. Pregnant women will receive monthly intensive dietary counseling, daily iron-folate, calcium supplementation, and at least four antenatal visits to local ANC service providers from enrollment before 16 weeks of gestation to delivery of the baby will be ensured.
  2. Adolescent girls will receive twice-monthly nutrition education sessions to improve dietary diversity scores from enrolment to 6 months of enrollment.
  3. Under 2y children will receive monthly growth monitoring and promotion, IYCF counseling
  4. Under 2y children for WASH counseling group will receive twice-monthly nutrition education sessions for 6months to improve maternal WASH practices
  5. Severely stunted children: Daily 1 egg for 3 consecutive months and 1 sachet of multiple micronutrient powder supplementation for 2 months.
  Interventions: Behavioral: Experimental - Intensive nutrition counselling for pregnant, adolescent and under2 children
- Control (No Intervention): Participants will receive the standard of care in the area

INTERVENTIONS:
Behavioral: Experimental - Intensive nutrition counselling for pregnant, adolescent and under2 children — Pregnant women: Intensive dietary counseling using diet chart for locally available food, and to attend antenatal care services from local ANC providers, daily Iron, folic acid, and calcium supplementation.
  Adolescent girls: Group sessions in the nutrition centers with the adolescent girls will be conducted twice monthly for 6 months. Iron and folic acid (200 mg ferrous fumarate and 400 μg folic acid); once weekly for 3 months; zinc 10 mg daily for 1 month.
  Children <2 years: Behavioral counseling sessions through monthly home visits on Infant and Young Child feeding, Growth monitoring and promotion, and water sanitation and hygiene, and food safety.
  Intensive WASH counselling: Intensive WASH counseling will be provided to separate group of child participants twice a month for 6 months.
  Severely stunted children: 1 egg supplementation for 3 months and 1 sachet of multiple micronutrient powder (1 RDA of vitamin A and C, iron-folic acid, and zinc) daily for 2 months.
  Other Names: Iron, folic acid and calcium supplementation for pregnant women; Zinc and iron-folate supplementation to adolescent gilrs; Egg supplementation to severely stunted children daily for 3 months to
  Arms: Experimental

SUMMARY:
The objective of the research project is to establish an evidence-based sustainable nutrition service delivery platform for optimizing pregnancy weight gain, increasing dietary diversity of adolescent girls, and ensuring proper physical growth of under 2 children.

Hypothesis

1. Pregnant Women: Intensive nutrition and WASH counseling, iron-folate, calcium supplementation during pregnancy, can improve gestational weight gain and improve hemoglobin status in pregnant women in a slum of Dhaka city
2. Adolescent girl: Iron and zinc supplementation and nutrition counseling on dietary diversity could improve nutritional status and dietary diversity score in adolescent girls of slums in Dhaka
3. Children <2 years: Counselling on IYCF, growth monitoring, and promotion, ensuring six-monthly vitamin A supplementation, counseling on WASH, treatment of acute malnutrition, and daily 1 egg supplementation for 3 months for severely stunted children can improve the nutritional status of children
4. Counselling to improve Water, Sanitation and Hygiene (WASH) practice: WASH intervention can improve EED biomarkers

DETAILED DESCRIPTION:
Background

1. Burden: The emergence of COVID-19 poses a substantial public health risk to the world. Our research done at the peak of the lockdown in Dhaka city showed that 90% of more than 200 households surveyed in a slum in Dhaka city and villages of Matlab in rural Bangladesh suffered from food insecurity, the situation was worse in the slum areas. Our previous work demonstrated that 50% of under-five children in slums have stunted growth, half of all children suffer from deficiency of zinc. Our recently completed study revealed that third-trimester weight gain was poor in general among rural women in Matlab, Bangladesh, and 54% of the women failed to gain adequate weight (>4 kg) in the third trimester.
2. Knowledge gap: Although the burden of undernutrition, as well as adverse consequences of nutritional impairment, is prominent in Bangladesh, there is no platform to implement sustainable nutrition delivery services in slums, particularly for children, adolescent girls, and mothers with pregnancy. In addition, there lack of data on the status of pregnancy weight gain, dietary diversity both in pregnant women and adolescent girls in slums. Evidence on the role of Infant and Young Child Feeding (IYCF), growth monitoring and promotion, micronutrient supplementation, and counseling on Water, Sanitation, and Hygiene (WASH) in improving childhood growth and ameliorating Environmental Enteric Dysfunction (EED) is also limited.
3. Relevance: Such lack of knowledge limits the success of nutritional programs being done in slums. Moreover, it is causing obstacles in reducing the nutritional burden among three vulnerable groups of the population.

Methods

This study will be conducted in the Bauniabadh and the adjacent slum areas of Dhaka city. This study includes a community survey, formative study, community-based nutrition intervention, and an evaluation of the programmatic intervention using a quasi-experimental design.

Bauniabadh slum area has a population of ~150,000. It has five blocks: A, B, C, D, and E. Blocks B, C, and E will be the intervention area for programmatic intervention and A and D will be the control area where no intervention will be provided. Blocks A, and D is separated from other blocks by a road, a school, and a water body.

At first, a community survey will be conducted to identify the total number of beneficiaries in both the control and intervention areas: under 2 years old children, adolescent girls, and pregnant women at or before 16 weeks of gestation.

The formative research includes 24-h dietary recalls, in-depth interviews with purposively selected household heads, women, adolescent girls, and focus group discussions with women and adolescent girls to explore the locally available foods to prepare nutritious diets for pregnant women and adolescent girls. Moreover, this formative study will help in tailoring the messages for group counseling sessions on nutrition and WASH on the perspectives of the slum dwellers in Dhaka city. All counseling materials for the programmatic intervention will be developed from data generated from the formative research and using existing materials.

In the intervention area, nutrition intervention will be provided to all pregnant women, adolescent girls, and children under the age of 2 years. For pregnant women, intensive dietary counseling will be provided through household visits. The intervention also includes daily iron-folate and calcium supplementation to the pregnant women for the remaining pregnancy period till childbirth, and at least four antenatal visits to local ANC service providers will be ensured. For all adolescent girls, monthly two nutrition education sessions for six months will be organized to improve dietary diversity. Adolescent girls will also receive weekly iron and folate supplementation for 3 months and 10 mg of zinc sulfate tablet daily for 1 month. Training research staff will do monthly growth monitoring and promotion for all under 2-year-old children. All children suffering from acute malnutrition will be treated and severely stunted children will be supplemented with one egg daily for 3 consecutive months and multiple micronutrient powders for 2 months. Additionally, counseling on water sanitation and hygiene, and food safety will be provided to the mother of the child participants. This program will also ensure community participation to improve the garbage disposal system, water supply and cleaning of drains in the area.

The primary outcome measures will be total pregnancy weight gain (kg) and rate of weight gain (kg/week) for pregnant women. Change in dietary diversity scores in adolescent girls, change in maternal WASH practices, and change in length-for-age z-score for children under the age of 2 years.

Evaluation will be done using a quasi-experimental design. Data related to outcome indicators will be collected from target groups from both the intervention and the controls areas.

At the end of the intervention, based on calculated sample sizes to see the changes in outcome variables, at a 5% level of significance with 90% power, we will need to enroll at least 199 pregnant women, 572 adolescent girls, 420 children below 2years, 89 children below 2years (WASH group) in each group. Based on previous data, we assume that the total available sample sizes for the programmatic intervention will be 400 pregnant women, 1200 adolescent girls, 1500 for children below 2years, and 178 children below 2years for WASH group. Therefore, our sample size will have more than enough power to test our hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women:

  * Age 18-39 years
  * Before 16 weeks of gestation
  * BMI 15-24.99 kg/m2 measured on enrolment
  * Have the plan to stay in the study area till delivery
  * Willing to participate in the study
  * Not enrolled in any nutrition project/programme currently

Adolescent girls:

* Aged 11-19 years
* Willing to participate in the study
* Not involved in any nutrition project/programme
* Will stay in the study area for the next 2 years

Children:

* Aged 0-24 months
* Youngest child of the household
* Caregivers have the plan to stay in the study area at least up to two years of age
* Not enrolled in any nutrition project/programme currently

Exclusion Criteria:

* Pregnant women:

  * Subject not willing to provide consent
  * Subject has the plan to migrate outside of the study area during the study period
  * Subject has a plan to go elsewhere ( village/ parents' house) for delivery
  * Any reported/diagnosed chronic diseases (such as hypertension, heart disease, chronic obstructive pulmonary disease, chronic kidney disease, chronic liver disease, pancreatic diseases, diabetes mellitus, thyroid dysfunction, immunological diseases, malignancy, or any other diseases which could impede compliance with the study protocol)
  * Extremely obese
  * Subject involved in any nutrition programme/ intervention currently

Adolescent girls:

* Subject not willing to give assent/consent
* Subject has the plan to migrate outside the study area during the study period
* Subject involved in any nutrition programme/intervention currently

Children:

* Caregiver/guardian not willing to provide consent
* Have the plan to migrate outside of the study area during the study period
* Child with any congenital anomaly
* Subject involved in any nutrition programme/intervention currently

Ages: 1 Day to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3278 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain | From the 16th week of gestation to child birth
  Change in gestational weight gain and rate of weight gain in the pregnant woman
Dietary Diversity | 6 months
  Change in Dietary Diversity of Adolescent Girl
Improve linear growth | 1 year
  Change in length for age z-score of children less than 2 years
Improved maternal WASH practices | 6 months
  Improvement in maternal WASH practics will be assessed through use of safe water, handwashing practice during critical times, use of hygienic/ improved toilet using a structured questionnaire

SECONDARY OUTCOMES:
Hemoglobin level of adolescent girl | 6 months
  A change in hemoglobin level Adolescent Girl
IYCF indicators | 1 year
  A change in WHO's core IYCF indicators for Children <2 years

OTHER OUTCOMES:
Hemoglobin level of Pregnant woman | 16 week of pregnancy to child birth
  A change in hemoglobin level of Pregnant woman

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Mahfuz, MBBS, MPH, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Diseases Research, Bangladesh (icddr,b), Dhaka, Dhaka Division, Bangladesh